CLINICAL TRIAL: NCT01458782
Title: A Randomized Trial Comparing Autologous Chondrocyte Implantation Using Collagen Membrane (ACI-C) Versus (Autologous Matrix Induced Chondrogenesis) AMIC for Repair of Cartilage Defects in the Knee
Brief Title: ACI-C Versus AMIC. A Randomized Trial Comparing Two Methods for Repair of Cartilage Defects in the Knee
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of North Norway (Other)
Collaborators: University of Tromso (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011/1159-3
Record Dates: First submitted 2011-10-17; First posted 2011-10-25 (Estimated); Results first posted 2025-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-01

CONDITIONS: Osteochondritis Dissecans; Osteoarthritis; Cartilage Injury; Osteonecrosis
Keywords: Cartilage repair; Chondrocytes; Stemcells
MeSH Terms: conditions — Osteochondritis Dissecans; Osteoarthritis; Osteonecrosis

STUDY DESIGN:
Intervention Model Description: RCT, Two arms ACI-C and AMIC
Oversight: Data Monitoring Committee: No

ARMS (2):
- ACI-C (Active Comparator): Autologous chondrocyte implantation using collagen membrane (ChondroGide) Please see reference 1 and 2 for details regarding ACI. In this study we are using the collagen membrane instead of periosteum- the other details are exactly the same as in our previous RCT.
  Interventions: Procedure: Treatment of cartilage defects in the knee
- AMIC (Active Comparator): Autologous matrix induced chondrogenesis. Microfracture of the defect and covering using the collagen membrane (ChondroGide).
  Please see reference 3 for details regarding AMIC
  Interventions: Procedure: Treatment of cartilage defects in the knee

INTERVENTIONS:
Procedure: Treatment of cartilage defects in the knee — Two groups, either ACI or AMIC. ACI includes an arthroscopy for harvesting of cartilage 3-4 weeks prior to the open cartilage surgery. AMIC includes only open surgery at one setting.
  Other Names: Autologous chondrocyte implantation; Autologous matrix induced chondrogenesis

SUMMARY:
ACI-C versus AMIC: A controlled randomized trial comparing Autologous Chondrocyte Implantation ( ACI) and Autologous Matrix Induced Chondrogenesis (AMIC) for repair of cartilage defects in the knee.

Eighty patients (Forty in each group) having symptomatic cartilage defects in their knee are planned to include in this study.

Both techniques will use the ChondroGide membrane from Geistlich to cover the defects. ACI includes an arthroscopy to harvest cartilage for cell cultivation in our lab located in Tromso. 3-4 weeks later using a mini arthrotomy the cells will be implanted under the ChondroGide membrane.

The AMIC group will be listed for a mini arthrotomy, cleaning of the defect, microfracture and cover of the defect using the same ChondroGide membrane.

In both groups stitches and fibrin glue will be used to fix the membrane.

Inclusion criteria:

Age between 18-60, Informed consent signed by patient, Symptomatic cartilage defect. Size more than 2 square cm.

Exclusion criteria Alcohol or drug abuse during the last three years, Inflammatory joint disease, Serious illness

Preoperative examination and follow up: Clinical examination and registration of KOOS (a validated knee score), VAS (visual analog pain scale) and Lysholm knee score. Radiographs of the involved knee including weightbearing standing radiographs of both knees. Kellgren- Lawrence classification will be used for grading of OA.

Patients will be checked after 1, 2, 5 and 10 years following surgery. Symptomatic patients having a new cartilage resurfacing operation or prosthesis will be listed as failures of the initial treatment.

Hypothesis: AMIC will be equal to ACI, and if that is the case this would be a benefit for the patients and the society. AMIC is much cheaper compared to ACI (needing an expensive cell cultivation and two surgeries).

Data will be analyzed using the SPSS statistical package.

DETAILED DESCRIPTION:
Please see referenced articles (1-3) for details regarding ACI and AMIC

ELIGIBILITY:
Inclusion Criteria:

* age between 18-60 yrs
* informed consent signed by patient
* symptomatic cartilage defect in the knee > 2 square cm

Exclusion Criteria:

* alcohol or drug abuse during the last three yrs
* inflammatory joint disease
* serious illness

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2011-10 (Actual); Primary Completion 2016-12-15 (Actual); Study Completion 2025-12-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Gunnar Knutsen, MD, PhD, Principal Investigator — University Hospital of North Norway; Ann Kristin Hansen, MD, PhD, Study Director — University Hospital of North Norway
Locations (1):
- University Hospital of North Norway, Tromsø, Troms, Norway

REFERENCES:
- [Background] Knutsen G, Drogset JO, Engebretsen L, Grontvedt T, Isaksen V, Ludvigsen TC, Roberts S, Solheim E, Strand T, Johansen O. A randomized trial comparing autologous chondrocyte implantation with microfracture. Findings at five years. J Bone Joint Surg Am. 2007 Oct;89(10):2105-12. doi: 10.2106/JBJS.G.00003. PMID 17908884
- [Background] Knutsen G, Engebretsen L, Ludvigsen TC, Drogset JO, Grontvedt T, Solheim E, Strand T, Roberts S, Isaksen V, Johansen O. Autologous chondrocyte implantation compared with microfracture in the knee. A randomized trial. J Bone Joint Surg Am. 2004 Mar;86(3):455-64. doi: 10.2106/00004623-200403000-00001. PMID 14996869
- [Background] Benthien JP, Behrens P. The treatment of chondral and osteochondral defects of the knee with autologous matrix-induced chondrogenesis (AMIC): method description and recent developments. Knee Surg Sports Traumatol Arthrosc. 2011 Aug;19(8):1316-9. doi: 10.1007/s00167-010-1356-1. Epub 2011 Jan 14. PMID 21234543
- [Derived] Fossum V, Hansen AK, Wilsgaard T, Knutsen G. Collagen-Covered Autologous Chondrocyte Implantation Versus Autologous Matrix-Induced Chondrogenesis: A Randomized Trial Comparing 2 Methods for Repair of Cartilage Defects of the Knee. Orthop J Sports Med. 2019 Sep 17;7(9):2325967119868212. doi: 10.1177/2325967119868212. eCollection 2019 Sep. PMID 31555714

RESULTS

PARTICIPANT FLOW:
Groups:
- AMIC: Autologous matrix induced chondrogenesis. Microfracture of the defect and covering using the collagen membrane (ChondroGide).
  Please see reference 3 for details regarding AMIC
  Treatment of cartilage defects in the knee: Two groups, either ACI or AMIC. ACI includes an arthroscopy for harvesting of cartilage 3-4 weeks prior to the open cartilage surgery. AMIC includes only open surgery at one setting.
Period: Overall Study
Arm/Group | ACI-C | AMIC
Started | 21 | 20
Completed | 21 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ACI-C | AMIC | Total
Number analyzed (Participants) | 21 | 20 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 20 | 41
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 37 (10.8) | 38 (8.2) | 37.5 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 12 | 19
  Male | 14 | 8 | 22
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Norway | 21 | 20 | 41

OUTCOME MEASURES:

1. Primary Outcome: Comparison Between the Two Groups of Mean Change From Baseline in Knee Injury and Osteoarthritis Outcome Score Total (KOOS) at Two Years.
Description: KOOS is a knee-specific instrument, developed to assess the patients opinion about their knee and associated problems. It holds 42 items in 5 sub-scales (pain, other symptoms, function in daily living, function in sport and recreation and knee-related quality of life). The questionnaire yields a total score ranging from 0-100. A higher score indicates better knee function. The reported number is the mean change in KOOS total score from baseline after two years for each group. A positive number represents an improved knee function score.
Time Frame: 2-years follow-up.
Population: Comparison between groups were performed on the intention-to-treat population (ITT)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ACI-C | AMIC
Number analyzed (Participants) | 21 | 20
score on a scale | 10.3 (16.0) | 18.1 (19.4)

2. Primary Outcome: Comparison Between the Two Groups of Mean Change From Baseline in Knee Injury and Osteoarthritis Outcome Score Total (KOOS) at Five Years.
Description: as for outcome 1
Time Frame: 5-years follow-up
Reporting Status: Not Posted, anticipated posting 2025-07

3. Secondary Outcome: Comparison Between the Two Groups of Mean Change From Baseline in Lysholm Score at Two Years.
Description: The Lysholm score is a scoring system for evaluating knee specific symptoms ranging from 0-100. Higher number indicates better knee function. The reported number is the mean change from baseline after two years for each group.
Time Frame: 2-years follow-up.
Population: Comparison between groups were performed on the intention-to-treat population (ITT).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ACI-C | AMIC
Number analyzed (Participants) | 21 | 20
score on a scale | 17.0 (14.9) | 19.7 (22.9)

4. Secondary Outcome: Comparison Between the Two Groups of Mean Change From Baseline in a Visual Analogue Scale (VAS) Pain Score at Two Years.
Description: The VAS scores describes the patients pain on a scale (0-100). Lower numbers, means less pain. The reported number is the mean change from baseline after two years for each group. Higher numbers represent more relief of pain.
Time Frame: 2-years follow-up.
Population: Intention to treat population (ITT)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ACI-C | AMIC
Number analyzed (Participants) | 21 | 20
units on a scale | 19.6 (25.9) | 30.6 (26.0)

5. Secondary Outcome: Failure
Description: Treatment failures were reported as either a "hard failure" or a "clinical failure." A hard failure was defined as the patients needing a new resurfacing procedure of the index lesion or implantation of a knee prosthesis. A clinical failure was defined as any deterioration in KOOS scores at 2-year follow-up compared to baseline. Diagnostic re-arthroscopy or arthroscopy with debridement of synovia or the defect was not considered a failure. Sum of "hard" and "clinical" failures at two years in each group are reported.
Time Frame: 2-years follow-up
Population: Intention to treat population (ITT)
Measure: Count of Participants; unit: Participants
Arm/Group | ACI-C | AMIC
Number analyzed (Participants) | 21 | 20
Participants | 3 | 5

6. Secondary Outcome: Comparison Between the Two Groups of Mean Change From Baseline in Lysholm Score at Five Years.
Description: The Lysholm score is a scoring system for evaluating knee specific symptoms ranging from 0-100. Higher number indicates better knee function. The reported number is the mean change from baseline after five years for each group.
Time Frame: Five-year follow-up
Reporting Status: Not Posted, anticipated posting 2025-07

7. Secondary Outcome: Comparison Between the Two Groups of Mean Change From Baseline in a Visual Analogue Scale (VAS) Pain Score at Five Years
Description: as for outcome 4
Time Frame: Five-years follow-up.
Reporting Status: Not Posted, anticipated posting 2025-07

8. Secondary Outcome: Failure
Description: Treatment failures were reported as either a "hard failure" or a "clinical failure." A hard failure was defined as the patients needing a new resurfacing procedure of the index lesion or implantation of a knee prosthesis. A clinical failure was defined as any deterioration in KOOS scores at 5-year follow-up compared to baseline. Diagnostic re-arthroscopy or arthroscopy with debridement of synovia or the defect was not considered a failure. Sum of "hard" and "clinical" failures at two years in each group are reported.
Time Frame: 5-years follow-up
Reporting Status: Not Posted, anticipated posting 2025-07

9. Secondary Outcome: Kellgren-Lawrence Baseline vs 5-years in Each Group
Description: Standing X-ray Rosenberg view of the knee obtained at baseline and 5-years follow up. X-rays were evaluated using the Kellgren-Lawrence scale by an independent orthopaedic surgeon.
Time Frame: 5-year follow-up
Reporting Status: Not Posted, anticipated posting 2025-07

ADVERSE EVENTS:
Time Frame: 2 years reported. 5 years will be reported later.
Description: No dedicated reporting system for adverse events, but the patients were followed up in such a manner that adverse events like death, surgical complications and re-operations would be reported.
Arm/Group | ACI-C | AMIC
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/20
Other Adverse Events (participants affected / at risk) | 3/21 | 3/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ACI-C (N=21) | AMIC (N=20)
Re-arthroscopy within 2 years (Musculoskeletal and connective tissue disorders) | 3 (4) | 3 (4) — One patient in each group had two rearthroscopies performed within the first two years after index surgery, thus three patients affected in each group, and a total of four events in each group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes